CLINICAL TRIAL: NCT05696262
Title: Effects of 6-minute Walking Exercise in Advanced Cancer and Non-cancer Patients: a Randomized Controlled Trial
Brief Title: 6 Minutes Walking Program for Terminally Ill Patients at Home or in an Institution
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Tsai-Wei Huang, professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: N202207044
Record Dates: First submitted 2022-11-15; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Walking Intervention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 6-walking program (Experimental): Perform 6 minutes of walking exercise 3 times a day, 3 days a week, in a comfortable manner.
  Interventions: Behavioral: 6-walking program
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Behavioral: 6-walking program — Perform 6 minutes of walking exercise 3 times a day, 3 days a week, in a comfortable manner
  Arms: 6-walking program

SUMMARY:
This study was conducted with a single-blind, randomized control method for 120 participants, 60 in the regular care group and 60 in the exercise intervention group. Those who meet the admission criteria will be contacted by phone and explained the purpose of the study. After asking for and obtaining consent, those who are willing to sign the consent form will be divided into groups and go to the home with the home care worker for the study. A suitable space was arranged for a 6-minute explanation and demonstration of walking exercise and a structured questionnaire to be filled out by the participant (the Barr's scale, Koch's scale and cognitive function assessment in the basic data were filled out by the facilitator), and the facilitator accompanied the participant during the process, giving explanations for unclear points to facilitate the completion of the questionnaire and to achieve a valid questionnaire. A trained research assistant was responsible for recruiting cases and receiving a study number and corresponding group assignment. Stratified random assignment (1:1) was used to divide the exercise intervention group and the usual care group. The study was listed using a randomized use of replacement blocks (block size 4). The assignment sequence was only available to the program facilitator and was not known to the other staff. Interventional measures Routine care group: A primary care team of physicians and nurse practitioners visited at least once a month for: (1) an initial intake visit (60-90 minutes) to provide a holistic assessment of disease intensity and prognosis, psychological distress, and social support; (2) at least one home care visit per month (30-60 minutes); (3) a telephone (4) Provide caregivers with social software and telepresence to solve caregiving problems (5) Provide exercise diaries to record daily activities of daily living (including vital signs, mobility, and fatigue). Exercise intervention group: In addition to the regular care group model, the intervention measure: 6 minute walk test (6MWT) is the simplest and most cost effective way to assess exercise. Pre-intervention equipment: 6-minute walk exercise video, yardstick, distance marker cone, measuring tape, exercise diary, smart bracelet, all subjects were provided with 6-minute walk exercise video and related equipment by the facilitator at intake. Before the test: explain the pre and post-test precautions, demonstrate the correct way to perform the test, and inform the patient to perform the test in a comfortable manner. In addition, the case was asked to wear the bracelet 24 hours a day for 7 days a week to observe the sleep quality. During the intervention period, if a case has the following conditions, the principle of implementation is as follows: (1) if the case has good walking ability, the case will be reminded to comply with the intervention (or keep the original physical activity) through telephone care and exercise diary; (2) if the case is physically able to walk but has low willingness to perform the 6-minute walk due to various conditions, the case will be reminded by family members or followed up by the researcher by telephone to improve the implementation rate; (3) if the case has difficulty getting out of bed due to the progress of the disease or treatment factors. (3) Cases with difficulty in getting out of bed or at risk of falling due to the progress of the disease or treatment factors; (4) Cases using oxygen to walk for 6 minutes in the area of the oxygen nasal cannula and tubing; if there is a risk of falling or injury during the procedure, please stop all activities immediately and ask the caregiver to monitor the vital signs and notify the facilitator and home care provider. If the patient needs to be taken to the hospital for treatment, assist in contacting the ambulance and send to the nearest hospital or the hospital where the patient usually goes for treatment; the host will visit the hospital and understand the situation and fill in the abnormal events. Outcome measurement: The family, primary caregiver, and the case are instructed to correctly measure the number of laps, distance, time, and number of times to walk, and to give instructions. Outcome measures were collected by the co-facilitators at intake, month 1, month 2, month 3, and month 6, and all data and assessment scales were tracked.

ELIGIBILITY:
Inclusion Criteria:

1. advanced cancer (cancer stage III or IV)
2. terminal ill disease
3. aged >=20 years
4. ECOG stage 0-3
5. Life expectancy =< 12 months

Exclusion Criteria:

1. unable to have normal conversation due to illness.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-16 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Steps count | Change from Baseline post exercise 5 min
  exercise outcome using pedometer
Steps count | Change from Baseline at 6 month.
  exercise outcome using pedometer

SECONDARY OUTCOMES:
Depression--Patient Health Questionnaire (PHQ-9) | Change from Baseline post exercise 5 min
  The PHQ-9 is the depression module, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day). It has been validated for use in primary care. It is not a screening tool for depression but it is used to monitor the severity of depression and response to treatment. high score mean higher emotion distress.
Depression--Patient Health Questionnaire (PHQ-9) | Change from Baseline at 6 month.
  The PHQ-9 is the depression module, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day). It has been validated for use in primary care. It is not a screening tool for depression but it is used to monitor the severity of depression and response to treatment. high score mean higher emotion distress.
cancer fatigue--BFI | Change from Baseline post exercise 5 min
  severity of fatigue level; measurement tool: Brief Fatigue Index
cancer fatigue--BFI | Change from Baseline at 6 month.
  severity of fatigue level; measurement tool: Brief Fatigue Index
Quality of Life--EQ5D-5L | baseline and six month.
  a 5-digit number that describes the patient's health state. The score increase means good quality of life.
Symptom Assessment---Chinese version of the Edmonton Symptom Assessment System，C-ESAS | baseline
  The ESAS includes 11 symptoms: pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, sleep, well-being, shortness of breath, and other. It uses a 0-10 numerical scale: 0 shows the absence of a symptom, and 10 shows the worst experience of the symptom.
Symptom Assessment---Chinese version of the Edmonton Symptom Assessment System，C-ESAS | Change from Baseline at 6 month.
  The ESAS includes 11 symptoms: pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, sleep, well-being, shortness of breath, and other. It uses a 0-10 numerical scale: 0 shows the absence of a symptom, and 10 shows the worst experience of the symptom.
Smart bracelet_Heart rate variability (HRV) | Continue wear bracelet five days to record HRV data.
  HRV is the physiological phenomenon of the variation in the time interval between consecutive heartbeats in milliseconds. A normal, healthy heart does not tick evenly like a metronome, but instead, when looking at the milliseconds between heartbeats, there is constant variation.
Trial Outcome Index (TOI) | Change from Baseline post exercise 5 min
  TOI is a useful tool to assess the physical and functional effects of treatment in patients. The higher score means higher outcome.
Trial Outcome Index (TOI) | Change from Baseline at 6 month.
  TOI is a useful tool to assess the physical and functional effects of treatment in patients. The higher score means higher outcome.

IPD SHARING:
Plan to Share IPD: No